CLINICAL TRIAL: NCT07382622
Title: Effect of JointIQ on Joint Discomfort in Healthy Subjects: A Randomized, Double-blind Trial
Brief Title: Effect of JointIQ on Joint Discomfort in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CS2-24092
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Joint Discomfort
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astragaloside Group (Experimental): 200mg astragaloside
  Interventions: Dietary Supplement: Astragaloside
- Placebo Group (Placebo Comparator): 200mg maltodextrin
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Astragaloside — Participants in the Astragaloside Group will receive one astragaloside capsule orally once daily after meals for 12 weeks. The capsule contains the active compound astragaloside, a component of the traditional herb Astragalus. Participants will be asked to continue their usual diet and physical activity levels during the study.
  Arms: Astragaloside Group
Dietary Supplement: Maltodextrin (Placebo) — Participants in the Placebo Group will receive one maltodextrin capsule orally once daily after meals for 12 weeks. The capsule is identical in appearance to the astragaloside capsule but contains no active astragaloside. Participants will be asked to continue their usual diet and physical activity levels during the study.
  Arms: Placebo Group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effects of astragaloside supplementation on joint discomfort in healthy adults. The primary goal is to determine if daily intake of astragaloside can improve knee joint function and reduce discomfort over a 12-week period. Participants will be randomly assigned to receive either an astragaloside capsule or a placebo capsule once daily. Aim to see if those taking astragaloside experience better mobility and fewer joint-related symptoms compared to those in the placebo group.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind clinical trial is to investigate the efficacy of astragaloside supplementation in enhancing joint health and physical function among healthy individuals aged 20 to 70 years.

Study Design and Procedures: Participants will be randomized into two groups: the intervention group (astragaloside) and the control group (placebo). Each participant will be instructed to consume one capsule daily after a meal for 12 weeks.

The study aims to address the following objectives:

Physical Function Assessment: To evaluate changes in knee joint mobility and strength using the Single-Leg Step-Down (SLSD) test and Range of Motion (ROM) measurements.

Subjective Symptoms and Quality of Life: To assess improvements in knee-related symptoms through the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire.

Biological Markers: To analyze blood biomarkers related to joint health and systemic response.

Comparative analysis between the astragaloside and placebo groups will be conducted to determine the statistical significance of the supplement's impact on joint function and discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, aged 18 to 75 years, with a body mass index (BMI) of 18-30 kg/m².
* Actively participates in regular exercise, including but not limited to soccer, basketball, tennis, rugby, running, or cycling, and engages in at least two training sessions per week during the study period.
* Experiences pain ≥5 on a Visual Analog Scale (VAS) during the Single-Leg Step-Down (SLSD) test when performing 30 to 150 steps.
* Has experienced knee discomfort within the last 3 months during or after physical activity.

Exclusion Criteria:

* Participation in another clinical trial within 30 days prior to study enrollment.
* Uncontrolled diabetes or currently using insulin therapy.
* Current smokers.
* History of heart failure.
* Previous bilateral knee replacement surgery.
* Current use of prescription COX-2 inhibitors, chondroitin sulfate, glucosamine sulfate or hydrochloride, collagen, fish oil, or vitamin D supplements and unwilling to discontinue these during the study.
* Likely to be lost to follow-up, non-compliant, or requiring concomitant medication that may interfere with study outcomes.
* Received intra-articular treatment within 3 months prior to study start.
* Medical conditions that may interfere with study results, such as cancer, cardiovascular disease (e.g., stroke, myocardial infarction), pregnancy, or breastfeeding.
* Hip, spine, or foot injuries that could affect study outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in knee joint stability via SLSD test at 12 weeks. | From baseline to Week 12
  The SLSD test evaluates functional knee stability and lower extremity muscle strength. The examiner records the number of successful repetitions or a quality score based on trunk and limb alignment. Higher scores (or higher number of repetitions) indicate better functional stability and joint control.
Change from baseline in knee Range of Motion (ROM) at 12 weeks. | From baseline to Week 12
  Knee ROM measures the degree of flexion and extension using a universal goniometer. The measurement is recorded in degrees. An increase in the range of degrees indicates improved joint mobility.
Change from baseline in KOOS score at 12 weeks. | From baseline to Week 12
  The KOOS questionnaire consists of 5 subscales: Pain, Symptoms, Activities of Daily Living, Sport and Recreation Function, and Knee-related Quality of Life (QOL). Standardized answer options are given (5-point Likert scale). Each subscale score is calculated as a percentage from 0 to 100. A score of 100 represents no knee problems and 0 represents extreme knee problems; therefore, a higher score indicates better outcomes.

SECONDARY OUTCOMES:
Change from baseline in serum inflammatory cytokine levels at 12 weeks. | From baseline to Week 12
  This measure evaluates the systemic inflammatory response by analyzing the concentrations of Pro-inflammatory cytokines, including Interleukin-6 (IL-6), Interleukin-8 (IL-8), Interleukin-1 beta (IL-1b), and Macrophage Inflammatory Protein-1 alpha (MIP1a). Blood samples will be analyzed using Enzyme-Linked Immunosorbent Assay (ELISA). A decrease in these biomarker concentrations (measured in pg/mL) indicates a reduction in systemic or joint-related inflammation.
Change from baseline in cartilage turnover biomarkers at 12 weeks. | From baseline to Week 12
  This measure assesses the balance between cartilage degradation and synthesis.
  Degradation Markers: C-terminal telopeptide of type II collagen (CTX-II), Cartilage Oligomeric Matrix Protein (COMP), and Matrix Metalloproteinase-13 (MMP-13).
  Synthesis Markers: Type II collagen markers (COL2a, PIIPC, and PIINP). Samples will be analyzed via ELISA. Lower levels of degradation markers and stable or higher levels of synthesis markers indicate improved cartilage health and reduced joint tissue breakdown.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan